CLINICAL TRIAL: NCT03579303
Title: A Comparative Study of Homoeopathic Treatment Versus Integrated Approach of Homoeopathy and Yoga in the Treatment of Menstrual Disorders in Females With Polycystic Ovarian Syndrome.
Brief Title: Homoeopathy and Yoga in the Treatment of Menstrual Disorders in Females With Polycystic Ovarian Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fr Muller Homoeopathic Medical College (Other)
Responsible Party: Principal Investigator, Dr Anita Fernandes, Professor, Fr Muller Homoeopathic Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AJP123
Record Dates: First submitted 2018-06-06; First posted 2018-07-06 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Menstrual Disorders; Polycystic Ovary Syndrome
Keywords: Homoeopathy; Yoga
MeSH Terms: conditions — Menstruation Disturbances; Polycystic Ovary Syndrome | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Homoeopathic remedies in PCOS (Active Comparator): Homoeopathic treatment for menstrual disorders in females with PCOS
  Interventions: Other: Homoeopathic Remedies
- Homoeopathic remedies and yoga in PCOS (Active Comparator): Homoeopathic treatment integrated with yoga therapy for menstrual disorders in females with PCOS
  Interventions: Other: Homoeopathic Remedies

INTERVENTIONS:
Other: Homoeopathic Remedies — comparison between homoeopathic treatment and integrated approach of homoeopathy and yoga in menstrual disorders of females with PCOS
  Other Names: Homoeopathic remedies and yoga therapy

SUMMARY:
This study is undertaken to compare effectiveness of homoeopathic treatment versus integrated approach of homoeopathy and yoga in the treatment of menstrual disorders in females with Polycystic ovarian syndrome.

DETAILED DESCRIPTION:
Polycystic ovarian syndrome (PCOS) is a complex metabolic, endocrine and reproductive disorder affecting approximately 5-10% of the female population in developed countries. The developing countries like China and India, undergoing rapid nutritional transitions due to westernised diets and lifestyle also indicate similar prevalence (9.13%). Its prevalence among infertile women is 15%-20%. The aetiology of Polycystic ovarian syndrome remains unclear; however, several studies have suggested that Polycystic ovarian syndrome is X-linked dominant condition.Women with Polycystic ovarian syndrome have abnormalities in the metabolism of androgens and oestrogen and in the control of androgen production. High serum concentrations of androgenic hormones, such as testosterone, androstenedione, and dehydroepiandrosterone sulfate (DHEAS), may be encountered in these patients. However, individual variation is considerable, and a particular patient might have normal androgen levels.

Polycystic ovarian syndrome is also associated with peripheral insulin resistance and hyperinsulinemia, and obesity amplifies the degree of both abnormalities. Insulin resistance in Polycystic ovarian syndrome can be secondary to a post binding defect in insulin receptor signalling pathways, and elevated insulin levels may have gonadotropin-augmenting effects on ovarian function. In addition, insulin resistance in Polycystic ovarian syndrome has been associated with adiponectin, a hormone secreted by adipocytes that regulates lipid metabolism and glucose levels. Both lean and obese women with Polycystic ovarian syndrome have lower adiponectin levels than women without Polycystic ovarian syndrome .

An anovulation and elevated androgen level suggests that under the increased stimulatory effect of luteinizing hormone (LH) secreted by the anterior pituitary, stimulation of the ovarian theca cells is increased. In turn, these cells increase the production of androgens (eg, testosterone, androstenedione). Because of a decreased level of follicle-stimulating hormone (FSH) relative to LH, the ovarian granulosa cells cannot aromatize the androgens to estrogens, which lead to decreased estrogen levels and consequent anovulation. Growth hormone and insulin-like growth factor 1 may also augment the effect on ovarian functioning.

The clinical manifestation of Polycystic ovarian syndrome varies from a mild menstrual disorder to severe disturbance of reproductive and metabolic functions. Women with Polycystic ovarian syndrome are predisposed to type 2 diabetes or develop cardiovascular disease . Factors implicated in the low fertility in these patients include anovulation, increased risk of early miscarriage, and late obstetric complications.

The diagnostic criteria of the syndrome were revised by the Rotterdam European Society for Human Reproduction/American Society of Reproductive Medicine (ASRM), where the following criteria were established: oligo/amenorrhea, clinical and biochemical signs of hyperandrogenism, and sonographically confirmed Polycystic ovarian syndrome. . Diagnostic criteria for Rotterdam diagnosis of polycystic ovary syndrome

Two of the following three criteria are required:

* Oligo/Anovulation
* Hyperandrogenism
* Clinical (hirsutism or less commonly male pattern alopecia) or
* Biochemical (raised FAI or free testosterone)
* Polycystic ovaries on ultrasound Other aetiologies must be excluded such as congenital adrenal hyperplasia, androgen secreting tumours, Cushing syndrome, thyroid dysfunction and hyperprolactinaemia Sonographic features of Polycystic ovarian syndrome include the presence of 12 or more follicles in each ovary measuring 2-9 mm in diameter and/or increased ovarian volume (>10 mL). This is regardless of follicle distribution or ovarian stromal echogenicity. One ovary fulfilling this definition is sufficient to define Polycystic ovarian syndrome.

Hirsutism is often classified in terms of the distribution and degree of hair growth, such as through pictorial scales. The most widely recognized scoring method is the Ferriman-Gallwey scale.

The Ferriman-Gallwey scale for hirsutism. A score of 1 to 4 is given for nine areas of the body. A total score less than 8 is considered normal, a score of 8 to 15 indicates mild hirsutism, and a score greater than 15 indicates moderate or severe hirsutism. A score of 0 indicates absence of terminal hair.

In a Cochrane Database Systematic Review article, Treatment options for polycystic ovary syndrome, It's mentioned about Alternative medicine and Polycystic ovarian syndrome. Alternative medicine has been emerging as one of the commonly practiced medicines for different health problems. Alternative medicines include many modalities, such as kinesiology, herbalism, homeopathy, reflexology, acupressure, acupuncture, and massage therapy.

Homoeopathy can be defined as a system of drug therapeutics based on the law of similars.Polycystic ovarian syndrome has a specific set of problems which need an individualistic approach.The concept of individualization takes into consideration the total response of the individual to unfavourable environment. This total response is seen through signs and symptoms on three planes: emotional, intellectual and physical where the life force manifests itself.The teachings of Dr Samuel Hahnemann(founder of homoeopathy)-that the human being is a unit -mind, body and spirit and that these are so correlated as to act freely and without any impediment when the vital principle, the spirit like force or dynamis is in equilibrium; yet if this equilibrium of health be thrown out of balance by the dysfunction of one member the whole is affected to a greater or less degree.Homoeopathy is the dominant option to treat Polycystic Ovarian Syndrome. Homoeopathic approach towards management of Polycystic ovarian syndrome is constitutional taking into account the patient's physical symptoms along with their mental and genetic makeup that individualizes the person. Early intervention with Homoeopathy can assist in preventing further progress and hence deterioration caused by Polycystic ovarian syndrome .

Homoeopathic constitutional treatment will help balance hyperactivity of the glands, regulate hormonal balance, dissolve the cysts in the ovaries and force them to resume normal functioning. Homoeopathic medicines will not upset the balance of endocrine secretions ,for the similimum(indicated remedy) will fill the demands of the system in all its parts without stimulating too much those organs which have maintained a relatively secure balance, in other words our remedies affect directly the vital energy which in itself establishes equilibrium. All the homoeopathic polycrest remedies (deep acting with a wide sphere of action) will yield richly to our search for effective remedies in endocrine disorders.Hence, Homoeopathic medicines can restore hormonal balance, normal ovulation, menstrual cycles, and also eliminate the need for hormone therapies and surgery. This can significantly increase the chances of conception. The different expressions of this disease can be managed effectively, safely and gently with Homoeopathic remedies.

Homoeopathy works towards nature. All homeopathy medicines are proved in human beings. It is very refined. It comforts modern living. The medicines have no negative side-effects. They are safe, effective and easy to attain cure. By taking homoeopathy medicines, ovulation and regular menses can be attained in a natural way.

Yogic life style, a form of holistic mind-body medicine, is known to reduce stress and sympathetic tone. Recent randomized controlled trial found holistic yoga program for 12 weeks to be significantly better than physical exercise in reducing Anti-Mullerian Hormone, Luteinizing Hormone and Testosterone, Modified Ferriman and Gallway (mFG) score for hirsutism and improving menstrual frequencies in Polycystic ovarian syndrome patients. Yoga not only addresses the problems of Polycystic ovarian syndrome but is likely to prevent the long term complications such as Cardio-vascular diseases, diabetes.

Following yogic practices are found to be useful in Polycystic ovarian syndrome :

1. Physical postures (Asanas - 1 min each):

   1. Surya Namaskara (Sun Salutation) for 10 min [5 rounds];
   2. Prone asanas:

      * Cobra Pose (Bhujangasana),
      * Locust Pose (Salabhasana),
      * Bow Pose (Dhanurasana)
   3. Standing asanas:

      * Triangle Pose (Trikonasana),
      * Twisted Angle Pose (Parsva -konasana),
      * Spread Leg Intense Stretch (Prasarita padottanasana),
   4. Supine asanas -

      * Inverted Pose (Viparita Karni),
      * Shoulder Stand (Sarvangasana),
      * Plough Pose (Halasana);
   5. Sitting asanas

      * Sitting forward Stretch (Paschimottanasana),
      * Fixed angle Pose (Baddha- konasana),
      * Garland Pose (Malasana)
2. Breathing Techniques (Pranayama - 2 min each):

   * Sectional Breathing (Vibhagiya- Pranayama),
   * Forceful Exhalation (Kapalabhati),
   * Right Nostril Breathing (Suryanuloma Viloma) 2 min,
   * Alternate nostril breathing (Nadishuddhi)
3. Guided relaxation (Savasana) for 10 min
4. OM Meditation (OM Dhyana) for 10 min
5. Group Lecture: Lectures, in the form of cognitive restructuring based on the spiritual philosophy underlying yogic concepts, spiritual coping strategies.

Homoeopathic medicines and yoga therapy being holistic approaches might effectively treat the complexity of the symptomatology in Polycystic ovarian syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18-36years
* Females diagnosed with Polycystic ovarian syndrome according to Rotterdam criteria.
* Participants willing to adopt a healthy life style and regularly practice yoga (at least 30 minutes for 5 days a week).

Exclusion Criteria:

* Diabetes mellitus, Cushing's disease, hyper-prolactinemia
* Untreated hypo or hyperthyroidism
* Adrenal hyperplasia and adrenal tumour
* Ovarian tumour hyperthecosis
* History of intake of drugs aldactone/metformin or history of oral contraceptive pills (OCP) use or intake of drugs known to interfere with carbohydrate metabolism 4 weeks prior to enrolment pregnancy, breast feeding cases with any systemic disease.

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 84 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
To assess if the interventions can facilitate regular menstrual cycle. | 3yrs
  Assessment of regularity in menstrual cycles will be done during the patients monthly visits to the out patient department ,recording the last menstrual period and duration of menses through a questionnaire

SECONDARY OUTCOMES:
To assess reduction in hyperandrogenism | 3yrs
  Assessment of reduction in hyperandrogenism will be done by Ferriman-Gallwey scale for hirsutism (Ref-Ferriman DM, Gallwey JD. Clinical assessment of body hair growth in women. J ClinEndocrinol 1961:21:1440-1447).
  Assessment of serum testosterone levels before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Subramanya Pailoor, Ph.D., Study Chair — Central University of Kerala, Kasaragod,; Dr Prema D'Cunha, MD,DNB, Study Chair — Father Muller Medical college,Kankanady,Mangalore
Locations (1):
- Fr Muller Homoeopathic Medical College, Mangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available .
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available within 6 months of study completion.
Access Criteria: Data access request will be reviewed by a external independent review panel. Requester's will be required to sign a data assess agreement.
URL: http://bethesda.org

REFERENCES:
- [Result] Prapas N, Karkanaki A, Prapas I, Kalogiannidis I, Katsikis I, Panidis D. Genetics of polycystic ovary syndrome. Hippokratia. 2009 Oct;13(4):216-23. PMID 20011085
- [Result] Badawy A, Elnashar A. Treatment options for polycystic ovary syndrome. Int J Womens Health. 2011 Feb 8;3:25-35. doi: 10.2147/IJWH.S11304. PMID 21339935
- [Result] Bern MJ, Sturbaum CW, Karayalcin SS, Berschneider HM, Wachsman JT, Powell DW. Immune system control of rat and rabbit colonic electrolyte transport. Role of prostaglandins and enteric nervous system. J Clin Invest. 1989 Jun;83(6):1810-20. doi: 10.1172/JCI114086. PMID 2723060
- [Result] Nidhi R, Padmalatha V, Nagarathna R, Amritanshu R. Effects of a holistic yoga program on endocrine parameters in adolescents with polycystic ovarian syndrome: a randomized controlled trial. J Altern Complement Med. 2013 Feb;19(2):153-60. doi: 10.1089/acm.2011.0868. Epub 2012 Jul 18. PMID 22808940
- See also: Yoga Exercises for PCOS | PCOS Treatment — http://www.artofliving.org/in-en/yoga/yoga-for-women/yoga-for-pcos
- See also: Boyle J, Teede H J,Polycystic ovary syndrome An update :Volume 41, No.10, October 2012 Pages 752-756. — http://www.racgp.org.au/afp
- Available data/document: Individual Participant Data Set: 123 — http://bethesda.org?data-id=123 — De-identified data for primary and secondary outcome measures

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT03579303/Prot_SAP_ICF_000.pdf